CLINICAL TRIAL: NCT05620082
Title: The RELISH Study: A Prospective Observational Study to Assess Compliance and Palatability of foRtifiEd Porridge Compared to Standard LIquid-baSed Oral Nutritional Supplementation in Hospitalised Older Adults With Malnutrition
Brief Title: The RELISH Study: Compliance and Palatability of Oral Nutritional Supplements in Hospitalised Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RHM MED1921
Record Dates: First submitted 2022-11-01; First posted 2022-11-17 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition
Keywords: Malnutrition; Oral nutritional supplementation; Compliance; Palatability; Older adult
MeSH Terms: conditions — Malnutrition; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New fortified porridge, then drink-based control (Experimental): Participants will first be given a new fortified porridge (Adams Vital Nutrition Ltd. High Protein Oats, 157g, 230kcal, 15g protein) twice per day for the first 2 days, in addition to normal meals in-between breakfast and lunch, and after dinner. Then given a drink-based control supplement (125g, 306kcal, 18g protein) for the next 2 days.
  Interventions: Dietary Supplement: Standard liquid-based oral nutritional supplement; Dietary Supplement: Fortified porridge
- Health care professionals (No Intervention): Health care professionals working on the wards receiving the intervention, including nurses, dietetics team, and health care assistants were interviewed to explore acceptability of products.
- Drink-based control, then new fortified porridge (Experimental): Participants will be given an anonymous drink-based control supplement twice per day for the first 2 days, in addition to normal meals, in-between breakfast and lunch, and after dinner. Then given a new fortified porridge supplement (157g, 230kcal, 15g protein) for the next 2 days.
  Interventions: Dietary Supplement: Standard liquid-based oral nutritional supplement; Dietary Supplement: Fortified porridge

INTERVENTIONS:
Dietary Supplement: Standard liquid-based oral nutritional supplement — An anonymous ready-made drink supplement: 125g, 306kcal, 18.3g protein.
  Arms: Drink-based control, then new fortified porridge; New fortified porridge, then drink-based control
Dietary Supplement: Fortified porridge — Vital Daily High Protein Oats (Adams Vital Nutrition Ltd.): 157g, 230kcal, 15g protein.
  Arms: Drink-based control, then new fortified porridge; New fortified porridge, then drink-based control

SUMMARY:
The RELISH study will investigate a new oral nutritional supplement (fortified porridge) for older adults in hospital who are undernourished (i.e., have malnutrition). Malnutrition is a lack of nutritional intake that can lead to poor recovery from illness, increasing hospital length of stay, and elevating healthcare costs. 22% of hospitalised older adults are estimated to have malnutrition. Oral nutritional supplementation (ONS) is key in the management of malnutrition. ONS are energy and nutrient dense products designed to increase dietary intake when diet alone is insufficient to meet daily nutritional requirements. However, for the ONS to be effective they need to be palatable (i.e., taste good), so that patients consume them (i.e., have good compliance) to reap the benefits of extra calories and protein. Normally, hospital patients are offered liquid based ONS (sip feeds). However, previous research has pinpointed that 56% of older adults on geriatric wards did not like sip feeds. Hence, exploration of compliance to different ONS formats is an important research direction to maximise malnourished older adult's nutritional intake. Therefore, the current study aimed to investigate the compliance and palatability of novel fortified porridge compared to traditional sip-feeds in malnourished older adults in hospital.

DETAILED DESCRIPTION:
22% of hospitalised older adults are estimated to be in a state of malnutrition. Malnutrition, also known as undernutrition, is a lack of nutritional intake leading to decreased fat free mass and diminished physiological functioning. Malnutrition impairs patient recovery, increasing hospital length of stay and escalating healthcare costs. Therefore, the identification and management of malnutrition is a vital patient-centred outcome to enhance older adult's health and quality of life and to enable cost-effective treatment and care.

A key method to support individualised nutritional care of hospital in-patients is the use of oral nutritional supplementation (ONS). ONS are energy and nutrient dense products designed to increase dietary intake when diet alone is insufficient to meet daily nutritional requirements. Overall, research suggests favourable impacts of ONS on nutritional status and healthcare costs, while the impact on functional outcomes and mortality are more controversial. A burgeoning evidence base attests to the importance of considering acceptability and compliance of ONS on adequate intake and thus effectiveness of ONS in practice.

Patient compliance to ONS considers the relationship between the amount of ONS prescribed and the amount of ONS ingested and is important to maximise clinical and cost-effectiveness. Palatability refers to the hedonic (i.e., pleasantness) evaluation of sensory factors, such as taste and smell, leading to alterations in food or fluid consumption. Supplemental preference may be affected by a multitude of factors such as taste, colour, smell, after taste and texture. Typically, hospital patients are offered liquid based ONS (sip feeds). However, previous research has pinpointed that 56% of older adults on geriatric wards did not like sip feeds. Hence, exploration of compliance to different ONS formats is an important research direction to maximise malnourished older adult's nutritional intake.

Malnourished hospitalised older adults should be offered an improved range and provision of ONS to suit patient preferences and maximise intake. For instance, an attractive alternative strategy is the use of energy and protein-dense meals (via fortification) or snacks (supplementation), including fortified bread, protein-enriched main meals and between meal snacks, such as biscuits, yoghurt and ice cream. Yet this is an understudied area, with limited data investigating compliance to alternative ONS products compared to ready-made drinks in hospital, such as powdered ONS and snacks, or their clinical effectiveness. Therefore, the current study aimed to investigate the compliance and palatability of novel fortified porridge compared to traditional sip-feeds in malnourished hospitalised older adults.

Research questions include:

1. What are the compliance rates (% intake) of fortified porridge compared to standard liquid based ONS in malnourished hospitalised older adults?
2. What are the palatability ratings (e.g., taste) of fortified porridge compared to standard liquid based ONS in malnourished hospitalised older adults?
3. What is the acceptability of fortified porridge compared to standard liquid based ONS in malnourished hospitalised older adults, including facilitators and barriers to their use on medical wards?

A mixed methods randomised controlled crossover design will be conducted to determine compliance and palatability of fortified porridge in malnourished hospitalised older adults compared to a liquid-based control ONS. The acceptability of products will be assessed through qualitative interviews to explore patients and healthcare professionals' experiences and views of using the nutritional supplements. Participants will be prescribed ONS twice per day for 4 days, in addition to normal meals, in a crossover design. The products will be offered in-between breakfast and lunch, and after dinner to reduce the detrimental long period of calorie absence experienced overnight.

ELIGIBILITY:
Inclusion Criteria:

* Older adults ≥65 years
* Patients on University Hospital Southampton (UHS) acute medical wards
* Medium-high risk of malnutrition (MUST score 1-4)
* Able to provide written consent

Exclusion Criteria:

* Patients that have used ONS in previous month
* Receiving enteral or parental nutrition
* Patients with a MUST score >4 (severely malnourished)
* Patients with a BMI ≤15
* Patients with chronic liver disease, renal failure, dysphagia
* Patients who have had major surgery within the preceding month
* Patients with a terminal illness
* Patients receiving end of life care
* Patients unable to eat by mouth (Nil By Mouth [NBM])
* Patients who require alternative ONS as advised by dietetic support

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha J Meredith, PhD, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southanmpton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 469 patients were screened for eligibility between April 22, 2024 and December 13, 2024 on medicine for older people wards and orthogeriatric wards in Southampton General Hospital, UK.
Pre-assignment Details: 114 patients were aproached after screening, 29 consented and 27 were randomised. We aimed to recruit 50 participants to the trial. Recruitment proved very challenging and after extending the study recruitment period, improving our recruitment strategies, and reviewing eligibility criteria, we recruited 27 patients to the trial and 5 staff. This number was deemed appropriate to answer our main research questions.
Groups:
- Porridge Supplement, Then Drink-based Control: Participants first received a new porridge supplement twice per day for 2 days, and then the drink-based control supplement twice per day for 2 days.
- Drink-based Control Supplement, Then Porridge Supplement: Participants first consumed a drink-based control supplement twice per day for 2 days, and then the new porridge supplement twice per day for 2 days.
- Health Professionals: Health professionals including nurses, dieticians, dietetic assistants, and health care assistants were interviewed to explore product acceptability
Period: Overall Study
Arm/Group | Porridge Supplement, Then Drink-based Control | Drink-based Control Supplement, Then Porridge Supplement | Health Professionals
Started | 16 | 11 | 5
Completed | 13 | 7 | 5
Not Completed | 3 | 4 | 0
Not completed — Discharged before study end | 1 | 4 | 0
Not completed — Moved to a different ward | 1 | 0 | 0
Not completed — Feeling too unwell | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- New Porridge Supplement, Then Drink-Based Control: Participants were given a new porridge supplement twice per day for 2 days, in addition to normal meals, in-between breakfast and lunch, and after dinner. Then a drink-based control supplement was given twice per day for 2 days.
  Standard liquid-based oral nutritional supplement: An anonymous ready-made drink supplement: 125g, 306kcal, 18.3g protein.
  Fortified porridge: Vital Daily High Protein Oats (Adams Vital Nutrition Ltd.): 157g, 230kcal, 15g protein.
- Health Care Professionals: Health care professionals working on the wards receiving the intervention, including nurses, dietetics team, and health care assistants.
- Drink-based Control Supplement, Then New Porridge Supplement: Participants were given a drink-based control supplement twice per day for 2 days, in addition to normal meals, in-between breakfast and lunch, and after dinner. Then a a new porridge supplement was given twice per day for 2 days.
  Standard liquid-based oral nutritional supplement: An anonymous ready-made drink supplement: 125g, 306kcal, 18.3g protein.
  Fortified porridge: Vital Daily High Protein Oats (Adams Vital Nutrition Ltd.): 157g, 230kcal, 15g protein.
- Total: Total of all reporting groups
Arm/Group | New Porridge Supplement, Then Drink-Based Control | Health Care Professionals | Drink-based Control Supplement, Then New Porridge Supplement | Total
Number analyzed (Participants) | 16 | 5 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.5 (6.4) | 40.20 (9.95) | 79.9 (10.8) | 74.5 (17.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 7 | 22
  Male | 6 | 0 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 15 | 3 | 11 | 29
  Any other White background | 1 | 2 | 0 | 3
Marital status [Count of Participants; unit: Participants] — Population: This baseline characteristic was not measured for health professionals participating in interviews
  Participants
    number analyzed (Participants) | 16 | 0 | 11 | 27
    Divorced | 3 | 0 | 2 | 5
    Married | 8 | 0 | 5 | 13
    Widowed | 5 | 0 | 4 | 9
Care provision [Count of Participants; unit: Participants] — This baseline characteristic was not measured for health professionals participating in interviews Population: This baseline characteristic was not measured for health professionals participating in interviews
  Participants
    number analyzed (Participants) | 16 | 0 | 11 | 27
    No care | 12 | 0 | 9 | 21
    Formal provision | 2 | 0 | 1 | 3
    Informal provision | 2 | 0 | 1 | 3
Frailty classification [Count of Participants; unit: Participants] — The Program of Research to Integrate Services for the Maintenance of Autonomy (PRISMA-7) screening tool was used to characterise participants' frailty status. The questionnaire contains seven items with a positive score of three or more indicating frailty. Population: This baseline characteristic was not measured for health professionals participating in interviews
  Participants
    number analyzed (Participants) | 16 | 0 | 11 | 27
    Frail | 12 | 0 | 6 | 18
    Not Frail | 4 | 0 | 5 | 9
Risk of sarcopenia [Count of Participants; unit: Participants] — The Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls (SARC-F) questionnaire was used as a measure to assess for sarcopenia. It comprises five components: strength, assistance in walking, rise from a chair, climbing stairs and falls. The scores range from 0 to 10, with a score of equal to or greater than four being predictive of sarcopenia and poor outcome. Population: This baseline characteristic was not measured for health professionals participating in interviews
  Participants
    number analyzed (Participants) | 16 | 0 | 11 | 27
    Sarcopenia | 13 | 0 | 7 | 20
    No sarcopenia | 3 | 0 | 4 | 7
Appetite [Count of Participants; unit: Participants] — Appetite was measured using the Simplified Nutritional Appetite Questionnaire (SNAQ), which has been validated to predict weight loss in community dwelling older adults and used to predict poor health outcomes in hospitalised older people. SNAQ is a four-item tool assessing appetite, satiety, taste of food and number of meals per day. SNAQ has a maximum score of 20, with a score of ≤14 indicating poor appetite. Population: This baseline characteristic was not measured for health professionals participating in interviews
  Participants
    number analyzed (Participants) | 16 | 0 | 11 | 27
    Poor appetite, high risk malnutrition | 8 | 0 | 6 | 14
    Good appetite, low risk malnutrition | 8 | 0 | 5 | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: This baseline characteristic was not measured for health professionals participating in interviews
  kg/m^2
    number analyzed (Participants) | 16 | 0 | 11 | 27
    (all) | 24.18 (5.05) |  | 24 (4.8) | 24.1 (5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Mean Oral Nutritional Supplement Consumed Per Day (%)
Description: Compliance to oral nutritional supplementation. Leftovers will be weighed (g) using weighing scales (Seca Model 875 digital weighing scale).
Time Frame: Measured daily during the 4 day testing period
Population: Participants with missing data were excluded from analysis. Health professionals completed interviews only.
Measure: Median (Inter-Quartile Range); unit: percentage of supplement consumed
Groups:
- Porridge Supplement: Participants consumed a new porridge supplement twice per day for 2 days.
- Drink-based Control Supplement: Participants consumed standard drink-based supplement twice per day for 2 days
Arm/Group | Porridge Supplement | Drink-based Control Supplement | Health Professionals
Number analyzed (Participants) | 18 | 18 | 0
percentage of supplement consumed | 26.31 [10.23 to 48.02] | 66.8 [26.29 to 75.37] |
Statistical Analysis 1: Comparison: Porridge Supplement vs Drink-based Control Supplement; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Energy (kcal) Consumed
Description: The average amount of daily energy consumed for each nutritional supplement (kcal)
Time Frame: Measured daily during the 4 day testing period
Population: Participants with missing data were excluded from analysis. Health professionals completed interviews only.
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Porridge Supplement | Drink-based Control Supplement | Health Professionals
Number analyzed (Participants) | 18 | 18 | 0
kcal | 141.41 [63.13 to 249.32] | 450.69 [198.69 to 492.33] |
Statistical Analysis 1: Comparison: Porridge Supplement vs Drink-based Control Supplement; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Protein Intake (g)
Description: The average daily amount of protein consumed from nutritional supplements (g)
Time Frame: Measured daily during the 4 day testing period
Population: Participants with missing data were excluded from analysis. Health professionals completed interviews only.
Measure: Median (Inter-Quartile Range); unit: grams (g)
Arm/Group | Porridge Supplement | Drink-based Control Supplement | Health Professionals
Number analyzed (Participants) | 18 | 18 | 0
grams (g) | 9.09 [4.06 to 16.02] | 26.51 [11.69 to 28.96] |
Statistical Analysis 1: Comparison: Porridge Supplement vs Drink-based Control Supplement; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Palatability of Oral Nutritional Supplement
Description: Palatability ratings, including appearance, smell, taste, sweetness, texture, thickness, aftertaste, mouth feel, and overall likability were assessed with a 7-point hedonic Likert scale (7 = definitely like, 6 = moderately like, 5 = mildly like, 4 = neither like nor dislike, 3 = mildly dislike, 2 = moderately dislike, 1 = definitely dislike).
Time Frame: Measured at baseline
Population: Participants with missing data were excluded from analysis. Health professionals completed interviews only.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Porridge Supplement | Drink-based Control Supplement | Health Professionals
Number analyzed (Participants) | 24 | 24 | 0
units on a scale
  Appearance | 5 [4 to 6] | 6.5 [4 to 7] |
  Smell | 4 [4 to 5.25] | 5.5 [4 to 7] |
  Taste | 4 [2 to 6.25] | 6.5 [4.25 to 7] |
  Sweetness | 4 [3 to 7] | 4.5 [2.25 to 7] |
  Texture | 4 [2 to 6] | 6 [4 to 7] |
  Thickness | 5 [2.75 to 7] | 6 [4 to 7] |
  Aftertaste | 4 [2.75 to 5] | 4 [2.25 to 7] |
  Feeling in mouth | 4 [1.5 to 5] | 4 [3 to 7] |
  Future choice | 4 [1.75 to 6] | 6 [4 to 7] |
Statistical Analysis 1: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Appearance of supplements; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Smell of supplements between groups; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Taste of supplements; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Sweetness of supplements; Test type: Superiority; p = 0.70, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Texture of supplements; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Thickness of supplements; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing Aftertaste of supplements; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing 'Feeling in mouth' of supplements; Test type: Superiority; p = 0.45, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Porridge Supplement vs Drink-based Control Supplement; Comparing 'Future choice' of supplements; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Total Caloric Intake (kcal)
Description: Total energy intake will be assessed through completion of patient food charts, including estimated proportion of meals consumed. Food charts are a part of patients' standard care and will be completed by the nursing team.
Time Frame: Completed daily during the 4 day testing period and 2 days before testing (baseline).
Population: Participants with missing data were excluded from analysis. Health professionals completed interviews only.
Measure: Median (Inter-Quartile Range); unit: kcal
Groups:
- Baseline: The baseline consisted of two days of food diaries analysed before nutritional supplements began
Arm/Group | Porridge Supplement | Drink-based Control Supplement | Health Professionals | Baseline
Number analyzed (Participants) | 20 | 20 | 0 | 20
kcal | 790 [593 to 979.5] | 703.25 [580.31 to 931.25] |  | 534.25 [410.13 to 804.75]
Statistical Analysis 1: Comparison: Porridge Supplement vs Drink-based Control Supplement vs Baseline; Test type: Superiority; p = 0.004, Related samples Friedman's Two-Way ANOVA — Pairwise comparisons with Bonferroni correction revealed a significant increase in total daily energy intake from baseline to porridge timepoints (p<0.001)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- New Porridge Supplement: Participants were given a new porridge supplement twice per day for 2 days, in addition to normal meals, in-between breakfast and lunch, and after dinner (Adams Vital Nutrition Ltd. High Protein Oats, 157g, 230kcal, 15g protein).
- Drink-Based Control Supplement: Participants were given a drink-based supplement twice per day for 2 days, in addition to normal meals, in-between breakfast and lunch, and after dinner (125g, 306kcal, 18g protein).
Arm/Group | New Porridge Supplement | Health Care Professionals | Drink-Based Control Supplement
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/5 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/5 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/5 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT05620082/Prot_SAP_000.pdf